CLINICAL TRIAL: NCT04899453
Title: Combined Intravitreal Methotrexate and ZR (Zanubrutinib& Rituximab) Regimen Followed by Zanubrutinib Maintenance in Newly-diagnosed Primary Vitreoretinal Lymphoma
Brief Title: Intravitreal MTX and ZR Regimen in Newly Diagnosed PVRL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-007
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Primary Vitreoretinal Lymphoma
Keywords: intravitreal methotrexate injection; rituximab; Primary vitreoretinal lymphoma; zanubrutinib
MeSH Terms: interventions — Methotrexate; Rituximab; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib/rituximab & intravitreal MTX (Experimental): Experimental arm will be treated with rituximab plus zanubrutinib (ZR) regimen for 6 cycles and followed by zanubrutinib maintenance for 2 years, meanwhile, intravitreal methotrexate will be given as protocol during the 1st year of treatment.
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Methotrexate — 400ug intravitreal injection every week for 4 doses in the induction phase, every 2 weeks for 2 doses as consolidation, then every month for 10 doses
Drug: Rituximab — Rituximab 375mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 6 cycles will be prescribed as protocol
Drug: Zanubrutinib — 160mg Bid, oral. 21-day cycle for 6 cycles in the induction phase and for 2 years in the maintenance phase

SUMMARY:
This is a prospective single-arm phase II study, and the purpose of this study is to evaluate the efficiency of ZR regimen (rituximab & Zanubrutinib) combined with intravitreal methotrexate and followed by Zanubrutinib maintenance in newly-diagnosed primary intraocular lymphoma. Progression-free survival (PFS) of the cohort is the primary endpoint.

DETAILED DESCRIPTION:
All the patients will be treated with ZR regimen (Rituximab 375mg/m2 IV d1, Zanubrutinib 160mg Bid, 21 days per cycle) as induction regimen, meanwhile intravitreal methotrexate was given at a dose of 400ug for 16 doses. The response will be evaluated every 3 cycles. After 3 Cycles, patients who achieved complete remission (CR) or partial remission (PR) will receive 3 more cycles of ZR regimen. The patients with stable disease (SD) or progressed disease (PD) will withdraw from the trial and receive salvage regimens. After total 6 induction cycles, the investigators evaluate the efficiency again, the patients with CR or PR will go to Zanubrutinib maintenance for 2 years or until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion. And the patients with SD or PD will receive a salvage regimen. During following-up, surveillance ophthalmologic examination, and brain magnetic resonance imaging (MRI) scans can be performed every 3 months up to the first 2 years, followed by the doctor visit every 6 months up to 5 years or the disease relapses.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed primary vitreoretinal lymphoma
* ECOG≤2
* creatinine clearance rate (CCR) ≥ 60ml/h, according to Cockcroft-Gault
* Total bilirubin # 2 upper limits of normal, alanine aminotransferase#ALT# < 3 upper limits of normal
* Sign the Informed consent
* Women of childbearing potential must understand that the study medication could have a potential teratogenic risk. They should undergo complete contraception during the study period.
* Male subjects must agree to use condoms throughout study drug therapy.

Exclusion Criteria:

* primary central nervous system lymphoma involved eyes and brain
* systemic B cell lymphoma involved eyes
* Pre-existing uncontrolled active infection
* Clinical evidence of grade 3 or 4 heart failure as defined by the New York Heart Association criteria
* Pregnancy or active lactation
* Co-existing tumors
* HIV or HBV or HCV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
2 years progression-free survival | from the date of treatment to the subject finished his 2 years follow-up phase or the disease relapsed or the death due to lymphoma
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow up without relapsing

SECONDARY OUTCOMES:
overall response rate (ORR) | 4 weeks after the end of 6 cycles of induction (each cycle is 21 days)
  ORR was calculated by the proportion of patients who achieved complete remission and partial remission

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China